CLINICAL TRIAL: NCT05346809
Title: Randomized Phase 2 Trial of Isatuximab During Autologous Stem Cell Collection and Transplantation Period in Patients With Multiple Myeloma, Relapsed Hodgkin's and Non-Hodgkin's Lymphoma
Brief Title: Isatuximab During Stem Cell Collection and Transplant in Patients With Multiple Myeloma and Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Divaya Bhutani (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Divaya Bhutani, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAT7444
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma; Multiple Myeloma; Non-Hodgkin Lymphoma; Relapsed Hodgkin's Disease, Adult
Keywords: Stem cell transplant
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isatuximab and Standard Procedures (Experimental): Subjects will receive the study drug Isatuximab in addition to standard procedures for transplant
  Interventions: Drug: Isatuximab
- Standard procedures (Experimental): Subjects will receive standard procedures for transplant.
  Interventions: Other: Standard Procedures

INTERVENTIONS:
Drug: Isatuximab — Isatuximab in IV form 10 mg/kg doses
  Other Names: Sarclisa
  Arms: Isatuximab and Standard Procedures
Other: Standard Procedures — Standard procedures (standard of care) for transplant
  Arms: Standard procedures

SUMMARY:
The purpose of this study is to see if Isatuximab can alter the immune system in patients with multiple myeloma or lymphoma upon recovery from the autologous stem cell transplantation. The investigators will see if Isatuximab makes changes to the immune system so that upon recovery from the transplant, the immune system can fight the cancer. This study will have two arms. On one arm (control arm), participants will receive standard transplant procedures and on the other arm (experimental arm), participants will receive Isatuximab in addition to the standard transplant procedures. The assignment to these arms is done randomly (determined by chance, like flipping a coin) by a computer. Each participant will have about 66% chance of getting on the experimental arm and about 33% chance of getting on the control arm.

DETAILED DESCRIPTION:
Relapse post-autologous stem cell transplantation (ASCT) remains a major challenge in the treatment of multiple myeloma (MM) and Lymphoma. The immune reconstitution post-ASCT has a major impact on the outcomes of ASCT, however effective methods to improve upon immune reconstitution have not been developed and the use of novel immunomodulators remains relatively unexplored. In addition, numerous studies have demonstrated the profound impact of graft composition on transplant outcomes, but not a single prospective study has addressed this issue successfully. In this study, the investigators intend to test a novel double pronged method of changing the immune repertoire post ASCT by modifying graft composition and improving effector T cell recovery and function post ASCT. In this study, the investigators intend to generate new information on immune modulation post-ASCT. In addition, the CD38 antibodies have not been evaluated as therapy for B-cell non-Hodgkin Lymphoma (NHL). If this study shows significant immunomodulator activity of this approach, cluster of differentiation 38 (CD38) antibodies could be further evaluated in combination with ASCT in NHL.

ELIGIBILITY:
Inclusion Criteria:

1. Following diagnoses are eligible for inclusion in the study:

   A) Multiple Myeloma with ASCT used as consolidation after first line induction therapy or at first relapse.

   B) Relapsed/Refractory Hodgkin's disease

   C) Non-Hodgkin's Lymphomas as follows
   * Relapsed/Refractory Diffuse large B cell lymphoma
   * Relapsed/Refractory indolent or relapsed/refractory transformed indolent B cell lymphomas as consolidation after second line therapy
   * Mantle Cell lymphoma as consolidation after first-line therapy
   * Peripheral T cell lymphoma as consolidation after first-line therapy or at relapse or primary refractory disease
2. Patients undergoing first ASCT will be eligible for the study.
3. Any prior therapy for the malignancy except CD38 antibody within the last 12 months is allowed.
4. Age ≥18 years
5. Life expectancy of greater than 6 months.

Exclusion Criteria:

1. Previously exposure to a CD38 antibody during the last 12 months.
2. Participants who are receiving any other investigational agents concurrently or received any investigational agent within the last 8 weeks.
3. History of severe allergic reactions or anaphylaxis attributed to compounds of similar chemical or biologic composition to Isatuximab.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Pregnant and Lactating women
6. HIV-positive status due to increased risk of infection when treated with immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in the total lymphocyte count | Day 30
  Change in total lymphocyte count measured from blood sample

SECONDARY OUTCOMES:
Number of Adverse Events | Up to 1 year
  The number of adverse events recorded for participants using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Percentage of participants with absolute lymphocyte count >500 cells/microliter | Day 30
  Percentage of participants with an absolute lymphocyte count of >500 cells/microliter on Day 30 post transplant
CD8 and CD4 Subsets | Up to 1 year
  Immune cell phenotyping ( cluster of differentiation 8 (CD8) and cluster of differentiation 4 (CD4) subsets) in the peripheral blood using flow cytometry based analysis
Percentage of activated B and T regulatory cells | Up to 1 year
  Percentage of activated B and T regulatory cells in the peripheral blood
Percentage of activated helper and effector T cells | Up to 1 year
  Percentage of activated helper and effector T cells in the peripheral blood
Percentage of Natural Killer (NK) cells | Up to 1 year
  Percentage of NK cells in the peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Divaya Bhutani, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Columbia University, New York, New York